CLINICAL TRIAL: NCT07143942
Title: Effects of Kinesio Taping on Gait Biomechanics in Patellar Tendinopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2024797
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-08

CONDITIONS: Patellar Tendinopathy / Jumpers Knee; Kinesio Taping
Keywords: patellar tendinopathy; Kinesio taping; gait biomechanics
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT-EDF+I-type combined with exercise therapy group (Experimental)
  Interventions: Behavioral: Kinesio Taping; Behavioral: exercise therapy
- KT-I type combined with exercise therapy group (Active Comparator)
  Interventions: Behavioral: Kinesio Taping; Behavioral: exercise therapy

INTERVENTIONS:
Behavioral: Kinesio Taping — KT-EDF + I Taping Method: With the knee flexed at 60°, two mesh-shaped Kinesio Tape strips were applied with natural tension over the painful area of the patellar tendon. A "jellyfish"-shaped Kinesio Tape strip was then placed with natural tension at the center of the knee joint, aligning its central hole with the treatment area. A thin KT strip was wrapped clockwise around this assembly. Next, the center of an I-shaped tape strip was stretched to 50%-75% tension and applied horizontally over the painful region of the patellar tendon, covering one-third to one-half of the width of the inferior pole of the patella. The ends were secured without tension. Additionally, a "Y"-shaped muscle tape was applied to the gluteus medius, running from the muscle origin to its insertion point. After taping, patients were instructed to keep the tape in place for five days before replacement. The KT-EDF + I taping intervention was continued for a total of eight weeks.
  Arms: KT-EDF+I-type combined with exercise therapy group
Behavioral: Kinesio Taping — KT-I Taping Method: With the knee joint bent to 30°, an "I"-shaped muscle tape was applied horizontally over the painful area of the patellar tendon (from the center toward both sides) with 50%-75% tension. Subsequently, a "Y"-shaped muscle tape was applied to the gluteus medius, running from the muscle's origin to its insertion point.
  After taping, patients were instructed to leave the tape in place for five days before replacement. The KT-I taping intervention was continued for a total of eight weeks.
  Arms: KT-I type combined with exercise therapy group
Behavioral: exercise therapy — Phase 1 aims to control load and alleviate pain. It includes isometric quadriceps exercises, wall-supported double-legged squats (at 90 degrees of knee flexion), Spanish squats, vastus medialis training, single-leg hip bridges with the affected leg supported, as well as stretching of the quadriceps, hamstrings, and triceps surae.
  Phase 2 focuses on gradually increasing load and strengthening exercise intensity. This phase incorporates eccentric and progressive loading movements, such as single-leg squats on a 25° inclined surface, lunges, vastus medialis activation, step-ups, and resistance exercises for the gluteal muscles.
  Phase 3 is designed to enhance functional capacity and facilitate a gradual return to sport. It involves energy-storage activities like jumping, box jumps, and interval running, with progressive increases in jump height, running distance, and speed. Once all exercises can be completed without knee discomfort for 24 hours, sport-specific training may be gradually

SUMMARY:
This study employed two distinct Kinesio Taping (KT) methods to treat patients with Patellar Tendinopathy (PT). It aimed to compare the efficacy between combined KT-EDF (Epidermis-Dermis-Fascia, EDF) with KT-I taping (I Strip Ligament Correction) and KT-I taping alone in improving pain and function among individuals with patellar tendinopathy. Furthermore, specialized equipment was used to assess changes in gait biomechanics before and after the intervention. Finally, this study integrated gait biomechanical data, scale scores, and surface electromyography signals to elucidate the potential mechanisms through which the combination of KT-EDF and KT-I taping improves gait biomechanics and reduces pain, thereby offering new therapeutic strategies for managing patellar tendinopathy with KT.

DETAILED DESCRIPTION:
Patellar Tendinopathy (PT), commonly referred to as "jumper's knee", is a frequent overuse injury resulting from sustained or high-intensity loading on the patellar tendon. It is characterized by tissue degeneration and microscopic tearing of the tendon due to repetitive mechanical stress. The most common site of pain is the junction between the inferior pole of the patella and the tibial tuberosity. Tenderness may also be present throughout the entire patellar tendon region. Pain is often accompanied by swelling and is exacerbated by physical activity. PT not only exhibits high prevalence among athletic populations but also tends to manifest persistent symptoms. Pain typically occurs during quadriceps-dependent activities such as running, jumping, and squatting. Increased exercise intensity aggravates the pain, which adversely affects the patient's quality of life, impairs athletic performance, and leads to abnormal gait biomechanics.

Kinesio Taping (KT) is widely employed in musculoskeletal rehabilitation and sports injury prevention. Previous studies have indicated that the Kinesio Taping-I Strip Ligament Correction (KT-I) method, a specific KT technique, can reduce pressure at the patellar tendon insertion on the inferior patellar pole and provide external mechanical support to the tendon structure. However, evidence regarding its effectiveness in improving pain, strength, and functional outcomes in PT patients remains inconsistent. Thus, further investigation is warranted to examine whether alternative KT taping methods can simultaneously alleviate pain and correct abnormal biomechanics in individuals with PT.

Among various KT techniques, the Epidermis-Dermis-Fascia (EDF) method employs mesh- or jellyfish-shaped tapes applied with minimal or natural tension (5%-10%) over the affected area. This technique has demonstrated promising results in pain relief and swelling reduction within musculoskeletal rehabilitation contexts. Furthermore, while existing studies on KT for PT have primarily focused on outcomes such as pain, strength, jumping and squatting performance, balance, and joint mobility, there is a notable lack of research regarding its effects on abnormal gait biomechanics in this population.

To address these gaps, this study combined EDF taping with KT-I taping for the treatment of PT patients. Gait parameters, surface electromyography (sEMG) signals of key lower limb muscles, isokinetic strength measurements, pain scores, and VISA-P (Victorian Institute of Sports Assessment-Patellar) scores were collected before and after the intervention. The outcomes were compared with those obtained from PT patients treated with KT-I taping alone. This study aimed to investigate the potential benefits of combined KT-EDF and KT-I taping in improving pain and function in PT patients, with particular emphasis on gait biomechanical characteristics. The ultimate goal is to enhance patients' quality of life, reduce sports-related injuries, and provide new insights and clinical references for the application of KT in the management of PT.

ELIGIBILITY:
Inclusion Criteria:

* Doppler ultrasound examination reveals structural tendon changes and/or increased tendon vascularity, or magnetic resonance imaging shows abnormal changes in the patellar tendon area;
* The patient has positive tenderness when pressing vertically upward on the tibial tuberosity;
* The patient has positive knee extension resistance test and/or patellar tendon pain during the single-leg squat test;
* The VISA-P scale score is less than 80 points;
* There is no allergic reaction to kinesio taping.

Exclusion Criteria:

* History of knee joint trauma;
* History of knee joint surgery;
* Taking painkillers in the past 2 weeks;
* Other knee joint diseases, such as knee osteoarthritis, knee tumors,rheumatoid arthritis, tuberculosis, etc.;
* Allergic reaction to Kinesio taping.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-08-31 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Vicon 3D gait test | 50 minutes
  subjects wore athletic shorts, fully exposing the waist and the area below the mid-thigh. After reflective markers were attached, subjects familiarized themselves with the movement collection requirements and procedures according to the testing protocol. They stood in the center of the testing room with their feet shoulder-width apart and upper limbs resting naturally at their sides, maintaining the subtalar joint in a neutral position. A static test was conducted to collect reference data for defining the coordinate systems of the bone segments.
  Subsequently, participants performed walking, jogging, side-cutting, jumping, and single-leg balance tasks at a self-selected comfortable pace. Sufficient rest was provided between trials to prevent fatigue. Five valid trials were collected for each movement, and the average of three trials was used for analysis.
Isokinetic muscle strength testing | 40minutes
  The testing was conducted by the same examiner using an isokinetic dynamometer (Con-Trex MJ, Germany).The subject sat with the hip flexed approximately 85 degrees. The distal end of the dynamic rod was fixed proximal to the medial malleolus. The trunk, pelvis, and mid-thigh were fixed to prevent other parts from compensating when the thigh exerted force. The knee joint's axis of motion was determined with the lateral femoral condyle as the axis. Test angular velocities were 60°/s, 180°/s, and 300°/s concentrically and 60°/s eccentrically, with 3-5 repetitions of each for concentric/eccentric knee extension or flexion contraction (90-10 degrees). A pre-test warm-up of 2-3 submaximal reps was performed, followed by a 1-2 minute rest period between each angular velocity. The test angular velocity was 60°/s, with isokinetic eccentric knee extension (90-10 degrees) performed for 3-5 repetitions of submaximal warm-up to familiarize the movement, followed by 3-5 maximal repetitions.

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain and VISA-P Scale | 5 miuntes
  Visual Analogue Scale for Pain：The VAS scale is usually a horizontal or vertical line 10 cm long with "0" and "10" marked on both ends. "0" represents "no pain" and "10" represents "worst possible pain." VISA-P Scale：A patellar tendinopathy rating scale is a reliable indicator of severity and pain. The VISA-P scale covers three areas: symptoms, function, and mobility. It consists of eight questions with a maximum score of 100. The theoretical minimum score is 0, and higher scores indicate less severe pain.
Surface electromyography signal parameters | 40minutes
  While patients performed gait biomechanical tests such as running, jumping, and side-cutting using the Vicon 3D device, a US-made Delsys wireless surface electromyography (SEM) instrument was used to simultaneously measure and collect EMG signals from the subjects' lower limb muscles during gait. The sampling frequency was set to 1500 Hz.
Plantar pressure test | 20minutes
  The subjects walked barefoot on a footscan® pressure plate (RSscan, 2×0.4 m, 16,384 sensors) at a self-selected speed. The pressure plate was placed in the middle of a 30-m runway. Before the test, the subjects warmed up and became familiar with the barefoot walking procedure, and then took the test at a self-selected appropriate speed. If the heel did not touch the ground first during a test or the subject's walking speed differed from the average of their normal walking speed by more than 10%, the test was considered invalid and the subject was asked to retest. Five valid test data were collected from each foot for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Beijing Key Laboratory of Sports Injuries, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No